CLINICAL TRIAL: NCT06434025
Title: Effect of Combination of Intravenous Iron and SGLT2 Inhibitor on Ventricular Function and Myocardial Iron Content in Patients With Heart Failure and Iron Deficiency.
Brief Title: IV Iron and SGLT2 Inhibitor on Ventricular Function and Myocardial Iron Content in Heart Failure With Iron Deficiency
Acronym: COMBINED-HF
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Principal Investigator, Luis Beck Da Silva Neto, Professor of Medicine, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 78861724.0.0000.5327; 2023-0428 (Other: AGH-Use HCPA)
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure, Systolic; Iron Deficiencies
Keywords: heart failure; iron deficiency; SGLT2 inhibitor; intravenous iron; clinical trial
MeSH Terms: conditions — Heart Failure, Systolic; Iron Deficiencies; Heart Failure | interventions — ferric carboxymaltose; dapagliflozin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: HFrEF, LVEF <40%, SGLT2i naive, and iron deﬁciency. Assigned to receive:
  1. intravenous iron + SGLT2i;
  2. intravenous iron + placebo of SGLT2i;
  3. placebo of both therapies.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ferric carboxymaltose + SGLT2 inhibitor (Experimental): Patients will receive 2 vials of ferric carboxymaltose 500 mg (Ferinject® 500 mg, Vifor-Pharma) IV, once; and Dapagliflozin 10 mg PO, once a day, for 30 days.
  Interventions: Drug: Iron Carboxymaltose; Drug: Dapagliflozin 10mg Tab
- ferric carboxymaltose + placebo of SGLT2 inhibitor (Active Comparator): Patients will receive 2 vials of ferric carboxymaltose 500 mg (Ferinject® 500 mg, Vifor-Pharma) IV, once; and placebo PO, once a day, for 30 days.
  Interventions: Drug: Iron Carboxymaltose; Drug: Placebo of Dapagliflozin
- Placebo of ferric carboxymaltose and placebo of SGLT2 inhibitor (Placebo Comparator): Patients will receive 2 vials of placebo IV, once; and placebo PO, once a day, for 30 days.
  Interventions: Drug: Placebo of Iron Carboxymaltose; Drug: Placebo of Dapagliflozin

INTERVENTIONS:
Drug: Iron Carboxymaltose — Iron Carboxymaltose 500 mg. 2 vials administered IV.
  Other Names: Ferinject
  Arms: ferric carboxymaltose + SGLT2 inhibitor; ferric carboxymaltose + placebo of SGLT2 inhibitor
Drug: Dapagliflozin 10mg Tab — Dapagliflozin 10mg Tab, PO, onde a day.
  Other Names: Forxiga
  Arms: ferric carboxymaltose + SGLT2 inhibitor
Drug: Placebo of Iron Carboxymaltose — Solution Sodium Chloride 0,9% 100 ml, IV, once.
  Other Names: Saline
  Arms: Placebo of ferric carboxymaltose and placebo of SGLT2 inhibitor
Drug: Placebo of Dapagliflozin — Equal shape and appearance tab as the tab containing Dapagliflozin 10 mg
  Arms: Placebo of ferric carboxymaltose and placebo of SGLT2 inhibitor; ferric carboxymaltose + placebo of SGLT2 inhibitor

SUMMARY:
Background. Treatment with intravenous iron has been shown to improve symptoms, functional capacity, and quality of life in patients with heart failure with reduced ejection fraction (HFrEF) and iron deﬁciency. However, the mechanisms underlying these beneﬁcial eﬀects remain unknown. SGLT2i seem to alter hematocrit and other hematological markers or iron content.

This study aims to measure cardiac magnetic resonance changes in myocardial iron content and in left ventricular function after administration of intravenous iron with and without the concomitant use of SGLT2 inhibitor in patients with HFrEF and iron deﬁciency.

DETAILED DESCRIPTION:
Background. Treatment with intravenous iron has been shown to improve symptoms, functional capacity, and quality of life in patients with heart failure with reduced ejection fraction (HFrEF) and iron deﬁciency. However, the mechanisms underlying these beneﬁcial eﬀects remain unknown. SGLT2i seem to alter hematocrit and other hematological markers or iron content. This study aims to measure cardiac magnetic resonance changes in myocardial iron content after administration of intravenous iron and to assess changes in left ventricular function in patients with HFrEF and iron deﬁciency.

Methods. Ninety-nine outpatient with symptomatic HFrEF, left ventricular ejection fraction (LVEF) <40%, SGLT2i naive, and iron deﬁciency will be assigned, to receive intravenous iron + SGLT2i; or intravenous iron + placebo of SGLT2i; or placebo of both therapies for 30 days. Myocardial iron will be evaluated by T2-star (T2*) cardiac magnetic resonance (CMR) sequencing before intravenous iron infusion. After 30 days, all patients will be reassessed by T2* CMR sequencing. The primary endpoint will be changes in LVEF and myocardial iron content at 30 days. Secondary endpoints will include correlations of these changes with myocardial iron content, functional capacity, quality of life, and cardiac biomarkers.

Conclusions. This study will determine the eﬀect of ferric carboxymaltose and its combination with SGLT2i on LVEF and its relationship with measures of myocardial iron content, functional capacity, and biomarkers in HFrEF and iron deﬁciency.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or over;
2. Ejection fraction (EF) ≤40%, estimated by color Doppler echocardiography or CMR or radionuclide ventriculography;
3. Serum ferritin <100 µg/L or serum ferritin between 100 and 299 µg/L and transferrin saturation <20%;
4. Serum hemoglobin between 9.5 and 13.5 mg/dL;
5. Patients must be SGLT2 naive;
6. Informed consent form (ICF) signed.

Exclusion Criteria:

1. Kidney disease requiring dialysis or chronic kidney disease not requiring dialysis with an estimated glomerular ﬁltration rate <30 mL/min/1.73 m2 calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation;
2. Severe primary valve disease;
3. Acute coronary syndrome requiring cardiac surgery or coronary artery bypass surgery in the past 3 months;
4. Patients already being treated for some type of non-iron deﬁciency anemia;
5. Blood transfusion within 30 days prior to CMR examination;
6. Patients with a pacemaker, cardiac resynchronization therapy, or implantable defibrillator;
7. Diagnosis of hemochromatosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-05-24 (Estimated); Primary Completion 2026-05-24 (Estimated); Study Completion 2026-11-24 (Estimated)

PRIMARY OUTCOMES:
left ventricular function assessed (LVEF) by CMR. | 30 days
  LVEF assessed by Cardiac Magnetic Resonance

SECONDARY OUTCOMES:
Myocardial iron content assessed by T2* CMR | 30 days
  Myocardial iron content assessed by T2* CMR
myocardial strain assessed by T2* CMR | 30 days
  myocardial strain assessed by T2* CMR

OTHER OUTCOMES:
six minute walk test (6MWT) | 30 days
  distance walked in six minute walk test
NT-proBNP | 30 days
  NT-terminal pro-B-type natriuretic peptide (NT-proBNP) levels
MLHFQ | 30 days
  Quality of life assessed by the Minnesota Living with Heart Failure Questionnaire
Hepcidin | 30 days
  Serum Hepcidin levels
Reticulocyte hemoglobin content | 30 days
  Reticulocyte hemoglobin content
Transferrin soluble receptors | 30 days
  Transferrin soluble receptors
Glomerular filtration rate | 30 days
  Glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: LUIS BECK DA SILVA, MD ScD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No